CLINICAL TRIAL: NCT01464125
Title: Evaluation of Fosmidomycin and Azithromycin When Administered Concurrently to Adult Subjects With Acute Uncomplicated Plasmodium Falciparum Malaria
Brief Title: Fosmidomycin and Azithromycin for Acute Uncomplicated Plasmodium Falciparum Malaria (P. Malaria) in Adults
Acronym: JP011
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jomaa Pharma GmbH (Industry)
Collaborators: Mahidol University (Other); Thammasat University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JP011
Record Dates: First submitted 2009-10-26; First posted 2011-11-03 (Estimated); Last update posted 2011-11-03 (Estimated); Status verified 2011-10

CONDITIONS: Malaria
Keywords: Malaria; Plasmodium falciparum; acute uncomplicated
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — fosmidomycin; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fos-Azi (Experimental): Open label single arm concurrent administration of fosmidomycin and azithromycin.
  Interventions: Drug: Fosmidomycin; Drug: Azithromycin

INTERVENTIONS:
Drug: Fosmidomycin — Fosmidomycin sodium capsules 450 mg x 4 twelve-hourly for three days
Drug: Azithromycin — Azithromycin capsules 250 mg x 3 twelve-hourly for three days

SUMMARY:
The aim of this study is to evaluate the role of azithromycin as a possible combination partner for fosmidomycin to protect it from its susceptibility to recrudescent infections when used as monotherapy for acute Plasmodium falciparum malaria while retaining its excellent safety profile.

DETAILED DESCRIPTION:
The scientific rationale for the use of this combination is to inhibit the ability of the parasite to synthesise isoprenoids, as precursors of many essential compounds including sterols, carotenoids and ubiquinones. This is effected through blockade of the non-mevalonate pathway by fosmidomycin as a potent inhibitor of 1-deoxy-D-xylulose 5-phosphate reductoisomerase coupled with targeting of protein biosynthesis by azithromycin through binding to the 50S ribosomal subunit. This mode of action contrasts with the ability of the human host to utilise the mevalonate pathway for isoprenoid synthesis and accounts for the safety profiles of both drugs through the mechanism of selective toxicity. Moreover it affords protection against cross resistance with existing chemotherapeutic agents.

The dose of fosmidomycin, equivalent to 30mg/kg twice daily for three days, selected for evaluation in this proof of concept study is derived from the highest dose that was administered in the Phase I safety tolerance studies. While the recommended dose of azithromycin for the treatment of bacterial infections is 250mg daily for three days, higher doses of up to 1500mg daily for three days have been evaluated for the treatment of malaria, in combination with artesunate or quinine.

ELIGIBILITY:
Inclusion Criteria:

* male and female subjects aged 15 to 55 years
* body mass index ≥ 18.5kg/M2
* uncomplicated P falciparum malaria with acute manifestations
* asexual parasitaemia between 500uL and 100,000uL
* ability to tolerate oral therapy
* able to give informed signed consent

Exclusion Criteria:

* signs of severe malaria, according to WHO criteria
* body mass index ≤ 18.5 kg/M2
* pregnancy by history or by positive urine test
* lactation
* mixed plasmodial infection
* concomitant disease masking assessment of response, including diabetes, uncontrolled hypertension, heart failure, hepatic dysfunction (alanine-amino transferase > 150 U/L), renal impairment (creatinine > 125 umol/L or 3 mg/dl), haemoglobin < 8g/dl, white cell count > 12000/uL
* anti-malarial treatment within previous 28 days
* symptomatic AIDS

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2008-11; Primary Completion 2009-10 (Actual); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
day 28 cure rate of >95% | 12 months
  Efficacy of fosmidomycin and azithromycin when co-administered to adults with acute uncomplicated P.falciparum malaria.
  Day 7 cure rate and Day 28 cure rates will be calculated from the following ratio: Number of subjects with clearance of asexual parasitaemia within seven days of commencement of treatment, without subsequent recrudescence within 28 days divided by total number of evaluable subjects.
Safety and Tolerance | 12 months
  To determine the safety and tolerance of fosmidomycin and azothromycin when co-administered orally over three days. Safety and tolerability will be evaluated by the incidence, intensity, seriousness and relationship of new adverse event(s), and clinically relevant laboratory changes. The drug will be considered as safe if there are no serious adverse events attributable to the study drug.
Day 7 cure rate of 100% | 12 months
  Efficacy of fosmidomycin and azithromycin when co-administered to adults with acute uncomplicated P.falciparum malaria.
  Day 7 cure rate and Day 28 cure rates will be calculated from the following ratio: Number of subjects with clearance of asexual parasitaemia within seven days of commencement of treatment, without subsequent recrudescence within 28 days divided by total number of evaluable subjects.

SECONDARY OUTCOMES:
Blood samples at 0,1,2,3,4,6,8,12,14,18,24, 26,30,36,38,42,48,50,54,60,62,66,72,78,84,90,96,108,120,144.168.240 hours | 12 months
  pharmacokinetic profile. Full profiles of pharmacokinetic parameters including Cmax, Tmax, peak, trough, Vd, AUC, T1/2a, T1/2t, renal and total Cl will be derived.
PCR corrected cure rates | 12 months
  to differentiate between reinfections and recrudescence

CONTACTS AND LOCATIONS:
Overall Officials: Srivicha Krudsood, Prof, Principal Investigator — Mahidol University
Locations (1):
- Mahidol University, Bangkok, Thailand